CLINICAL TRIAL: NCT01258517
Title: The Effect of the Type and the Method of Surfactant Administration on Oxygenation in Preterm Infants: a Near Infrared Spectroscopy Study
Brief Title: The Effect of Surfactant Administration on Cerebral Oxygenation
Status: Suspended | Type: Observational
Why Stopped: principle investigator moved to an another hospital
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NIRS-018
Record Dates: First submitted 2010-12-07; First posted 2010-12-13 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2010-11

CONDITIONS: Respiratory Distress Syndrome; Prematurity
Keywords: RDS; surfactant; cerebral oxygenation; near infrared spectroscopy
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group 1, group 2, group 3, group 4: administration of beractant with single lumen ET tube administration of poractant with single lumen ET tube administration of beractant with double lumen ET tube administration of poractant with double lumen ET tube
  Interventions: Device: near infrared spectroscopy (INVOS 5100)

INTERVENTIONS:
Device: near infrared spectroscopy (INVOS 5100) — monitorization of cerebral oxygenation by INVOS 5100 during surfactant administration

SUMMARY:
The purpose of this study is to assess changes in cerebral oxygenation during two different types (beractant and poractant) and two different routes (double lumen or single lumen endotracheal tube) of surfactant administration using near infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of respiratory distress syndrome <32 gestational weeks and/or <1500 g birthweight

Exclusion Criteria:

major congenital anomalies complex congenital heart diseases

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: <32 week or <1500 g required surfactant treatment for established RDS
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
to determine the optimal and the most safe surfactant administration technique with regard to cerebral oxygenation as measured by near infrared spectroscopy in low birth weigh infants | up to 36 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Neonatal Intensive Care Unit, Ankara, Turkey (Türkiye)